CLINICAL TRIAL: NCT03078153
Title: The Effect of Social Media Support and Financial Incentives on Adherence to HIV Pre-exposure Prophylaxis in Young MSM of Color in Washington, DC
Brief Title: Effect of Social Media Support and Financial Incentives on PrEP Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Marc O. Siegel, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 111642; 1P30AI117970 (NIH)
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Pre-Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Financial Incentive (Experimental): Provided financial incentive at 3-month and 6-month follow-up visits
  Interventions: Behavioral: Financial Incentive
- Social Media Group (Experimental): Provided social media support through a facebook group for 6 months
  Interventions: Behavioral: Social Media Group
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Financial Incentive — Participants will receive a $50 gift card at 3- and 6- month follow-up visits.
  Arms: Financial Incentive
Behavioral: Social Media Group — Participants will be invited to a study Facebook group which will have links to PrEP information and provide a forum for participants to ask questions and communicate their experience with PrEP
  Arms: Social Media Group

SUMMARY:
The purpose of this study is to determine if social media support and financial incentives improve adherence to Truvada as PrEP in African American, Latino and Asian MSM aged 18 to 24 living in the Washington, DC area who are at high risk for HIV acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Male assigned at birth (regardless of current gender identity)
* Age 18-24
* Black/African American, Latino or Asian
* HIV negative
* History of unprotected anal sex with a man in the last 6 months
* Living within the DC metropolitan statistical area and anticipate remaining within the DC area for the next 6 months
* Not enrolled in any other HIV prevention trial
* Interested in taking PrEP
* Not a current PrEP user and have not taken PrEP in the last 30 days
* Able to provide informed consent

Exclusion Criteria:

* Female sex at birth
* Age younger than 18 or older than 24
* Caucasian
* HIV positive
* Actively taking PrEP or having taken PrEP within 30 days of enrollment
* Chronic hepatitis B infection
* Known renal insufficiency
* On probation or parole
* Any other conditions that the Principal Investigator may consider a contraindication to enrolling in the study

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male at birth (regardless of current gender identity)
Enrollment: 57 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Adherence To Truvada | 6 months
  Level of Truvada drug levels inside red blood cells (performed by dried blood spots)

SECONDARY OUTCOMES:
New Cases of HIV | 6 months
  Number of reactive HIV rapid and 4th generation tests
Incidence of STIs | 6 months
  Positive RPR, oropharyngeal/rectal/penile chlamydia and gonorrhea during study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Siegel, MD, Principal Investigator — The GW Medical Faculty Associates
Locations (1):
- The GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No